CLINICAL TRIAL: NCT05286684
Title: Feasibility of Exosome Analysis in Cerebrospinal Fluid During the Diagnostic Workup of Metastatic Meningitis From Breast Cancer
Brief Title: Feasibility of Exosome Analysis in Cerebrospinal Fluid During the Diagnostic Workup of Metastatic Meningitis
Acronym: Exo-LCR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Oscar Lambret (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Exo-LCR-1807
Record Dates: First submitted 2022-01-31; First posted 2022-03-18 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2024-11

CONDITIONS: Breast Cancer
Keywords: leptomeningeal metastases; proteomic profile; cerebrospinal fluid; cytology analysis
MeSH Terms: conditions — Breast Neoplasms; Meningeal Carcinomatosis | interventions — Referral and Consultation; Spinal Puncture

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Study process (Experimental): Consultation, Cerebral and medullary MRI, lumbar puncture, CSF sampling, blood sample, collection of breast fluid
  Interventions: Procedure: Consultation; Procedure: Cerebral and medullary MRI, lumbar puncture, CSF sampling; Biological: biological test

INTERVENTIONS:
Procedure: Consultation — History of the disease, anatomopathological and molecular biological data concerning the initial tumor; Collection of treatments received and/or in progress by the patient for her meningeal tumor (chemotherapy, targeted therapy, radiotherapy, surgery, corticosteroids, antiepileptics); Evaluation of the general condition and neurological status.
Procedure: Cerebral and medullary MRI, lumbar puncture, CSF sampling — diagnosis of leptomeningeal involvement
Biological: biological test — 5 ml of additional CSF after diagnostic lumbar puncture for proteomic analysis, 50-100 µl of breast aspiration fluid (NAF) for patients with an existing breast tumor, for proteomic analysis 10 ml of blood for proteomic analysis

SUMMARY:
The investigators are interested in one of the most frequent tumor types causing leptomeningeal metastasis in order to investigate whether a profile can be established by a high-throughput clinical proteomic approach. All the data acquired will allow a tailored and promising approach to improve the knowledge of metastatic tumor meningitis.

DETAILED DESCRIPTION:
The primary objective is to describe on an exploratory basis the association between the type of proteomic profile from cerebrospinal fluid (CSF) microvesicles (from unsupervised bioinformatics analysis) and CSF cytology analysis (positive, negative, equivocal) in breast cancer patients with suspected leptomeningeal metastases, on initial CSF samples (hereafter referred to as initial proteomic profile and initial cytology).

ELIGIBILITY:
Inclusion Criteria:

* Patient with histologically proven breast cancer;
* Patient with suspected metastatic leptomeningeal involvement;
* Age ≥ 18 ans ;
* WHO performance status ≤ 2 ;
* Affiliation to the National Social Security System ;
* With informed and signed consent

Exclusion Criteria:

* History of another cancer than the one for which the patient is referred;
* Contraindication to lumbar puncture or cerebrospinal MRI
* Pregnant or breastfeeding woman

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Breast cancer
Enrollment: 7 (Actual)
Dates: Start 2023-01-04 (Actual); Primary Completion 2023-11-15 (Actual); Study Completion 2023-11-15 (Actual)

PRIMARY OUTCOMES:
CSF protein composition | 36 months
  The CSF proteomic profile will be obtained by an unsupervised bioinformatics analysis of the CSF collected during the initial diagnostic workup for all patients and in case of renewal of the initial lumbar puncture if the 1st one was not exploitable for the CSF cytological analysis.
  The bioinformatics analysis will allow to obtain the protein composition and to establish proteomic profile.
cytological analysis of the CSF | 36 months
  The cytological analysis of the CSF will allow to obtain 3 possible results: Positive / Negative / Equivocal at the time of the initial diagnostic workup for all patients and in case of renewal of the initial LP if the 1st one was not exploitable for the cytological analysis of the CSF, for all patients.

CONTACTS AND LOCATIONS:
Overall Officials: Claire Cheymol, MD, Principal Investigator — Centre Oscar Lambret
Locations (1):
- Centre Oscar Lambret, Lille, Hauts-de-France, France

IPD SHARING:
Plan to Share IPD: No